CLINICAL TRIAL: NCT04865003
Title: Prognostic Factors for Descending Necrotizing Mediastinitis Development in Deep Space Neck Infections - A Retrospective Study
Brief Title: Prognostic Factors for Descending Necrotizing Mediastinitis Development in Deep Space Neck Infections
Status: Completed | Type: Observational
Sponsor: Clinical Center of Vojvodina (Other)
Responsible Party: Principal Investigator, Denis Brajković, Principal Investigator, Clinical Center of Vojvodina
Other Study IDs: 1208983
Record Dates: First submitted 2021-04-14; First posted 2021-04-29 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Infection; Mediastinitis; Neck Abscess; Inflammation
MeSH Terms: conditions — Infections; Mediastinitis; Inflammation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- DNI group: patients with infection of two or more deep neck spaces (DNI group)
  Interventions: Other: treatment of infection
- DNI + DNM group: patients with infection of two or more deep neck spaces with secondary descending necrotizing mediastinitis (DNI + DNM group)
  Interventions: Other: treatment of infection

INTERVENTIONS:
Other: treatment of infection

SUMMARY:
Descending necrotizing mediastinitis (DNM) is the most serious complication of deep neck infections (DNI) with high mortality. The objective of this retrospective study was to evaluate possible prognostic factors for DNM development in deep space neck infections.

DETAILED DESCRIPTION:
Descending necrotizing mediastinitis (DNM) is the most serious complication of deep neck infections (DNI) with high mortality. The objective of this retrospective study was to evaluate possible prognostic factors for DNM development in deep space neck infections. The study enrolled patients admitted to the Emergency Center of Vojvodina with the diagnosis of multispace DNI with or without DNM either as the primary diagnosis or with discharged diagnosis after surgical treatment during 7-years period. The data were obtained from patient medical records.

ELIGIBILITY:
Inclusion Criteria:

* patients admitted to the hospital due to deep neck infection affecting two or more spaces with or without descending necrotizing medioastinitis
* complete diagnosis and treatment data available from medical charts

Exclusion Criteria:

* incomplete medical data
* infection confined to one deep neck space
* patients treated under local anesthesia
* patients with superficial skin infections
* iatrogenic infections
* infected tumors

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: This study enrolled patients admitted to the Emergency Center of Vojvodina with the diagnosis of multispace DNI with or without DNM either as the primary diagnosis or with discharged diagnosis after surgical treatment.
  The diagnosis of DNM was based on standard Estrera et al. diagnostic criteria. Cases included in the study comprised patients admitted to the hospital due to DNI affecting two or more spaces with or without DNM. Cases were excluded from the study if complete medical data could not be obtained from medical charts.
Sampling Method: Non-Probability Sample
Enrollment: 289 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Incidence of mediastinitis | Within 6 hours of admission
  Neck and chest computed tomography (CT)

SECONDARY OUTCOMES:
Microbiological findings in DNI and DNM | Within 1 week of admission
  Prevalence of microorganisms in mediastinitis
Average number of hospital days | Through study completion, an average of one month
  Comparison of average number of hospital days in DNI and DNM
Incidence of complications | Within 30 days from admission
  Complications among DNI and DNI+DNM groups
Number of infected deep neck spaces | Within 6 hours of admission
  Neck and chest computed tomography (CT)

CONTACTS AND LOCATIONS:
Overall Officials: Aleksandar Kiralj, PhD, Study Director — Clinical Center of Vojvodina

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Prado-Calleros HM, Jimenez-Fuentes E, Jimenez-Escobar I. Descending necrotizing mediastinitis: Systematic review on its treatment in the last 6 years, 75 years after its description. Head Neck. 2016 Apr;38 Suppl 1:E2275-83. doi: 10.1002/hed.24183. Epub 2016 Feb 1. PMID 26829352
- [Result] Qu L, Xu H, Liang X, Cai X, Zhang W, Qian W. A Retrospective Cohort Study of Risk Factors for Descending Necrotizing Mediastinitis Caused by Multispace Infection in the Maxillofacial Region. J Oral Maxillofac Surg. 2020 Mar;78(3):386-393. doi: 10.1016/j.joms.2019.11.017. Epub 2019 Nov 26. PMID 31862339
- [Result] Sarna T, Sengupta T, Miloro M, Kolokythas A. Cervical necrotizing fasciitis with descending mediastinitis: literature review and case report. J Oral Maxillofac Surg. 2012 Jun;70(6):1342-50. doi: 10.1016/j.joms.2011.05.007. Epub 2011 Aug 6. PMID 21820786
- [Result] Boscolo-Rizzo P, Da Mosto MC. Submandibular space infection: a potentially lethal infection. Int J Infect Dis. 2009 May;13(3):327-33. doi: 10.1016/j.ijid.2008.07.007. Epub 2008 Oct 25. PMID 18952475
- [Result] Kimura A, Miyamoto S, Yamashita T. Clinical predictors of descending necrotizing mediastinitis after deep neck infections. Laryngoscope. 2020 Nov;130(11):E567-E572. doi: 10.1002/lary.28406. Epub 2019 Nov 20. PMID 31747058
- [Derived] Brajkovic D, Zjalic S, Kiralj A. Prognostic factors for descending necrotizing mediastinitis development in deep space neck infections-a retrospective study. Eur Arch Otorhinolaryngol. 2022 May;279(5):2641-2649. doi: 10.1007/s00405-021-07081-0. Epub 2021 Sep 20. PMID 34542654